CLINICAL TRIAL: NCT07250425
Title: Development of a Novel, Cost-Effective Gait Training Device Utilized at Home for the Neurological Patient Population
Brief Title: Development and Efficacy of a Novel, Cost-Effective Gait Training Device Utilized at Home for Stroke Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Healing Innovations (Other)
Collaborators: Kessler Foundation (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Julie Hartman, Doctor of Physical Therapy, Vice President of Clinical Development & Strategy, Healing Innovations
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R44HD113451 (NIH); 1R44HD113451-01A1 (NIH)
Record Dates: First submitted 2025-05-28; First posted 2025-11-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Neurological Diseases or Conditions; Hemiparesis;Poststroke/CVA; Gait Disorders, Neurologic; Post Stroke Fatigue; Motor Recovery; Walking Difficulty; Balance Impairment; Falls Prevention; Hemiparesis; Mobility Limitation
Keywords: in-home rehabilitation; Robotic-Assisted Gait Training; gait training device; stroke recovery; functional mobility; rehabilitation technology; remote monitoring; rehabilitation robotics; Fitbit Step Tracking; Self-Directed Gait Training; high-intensity gait training; Neurorehabilitation Research; Lower Limb Rehabilitation; Motor Function Recovery; Physical Therapy; Walking Endurance; task specific walking practice; neurological recovery; stroke rehabilitation; home exercise program; Rise&Walk InHome; daily step count; 6-minute walk test; 10-meter walk test
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Mobility Limitation; Paresis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either home-based robotic gait training with the Rise&Walk InHome device plus usual care or usual care alone for 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Group: Rise&Walk InHome Walking Group (Active Comparator): Participants will receive an in-home Rise&Walk InHome robotic gait training device in addition to their usual rehabilitation care. They will be instructed to perform 30-minute sessions of device-based walking four times per week for 12 weeks, with individualized device parameters and weekly remote check-in calls with the study team to monitor safety, adherence, and progression.
  Interventions: Device: Rise&Walk InHome by Healing Innovations
- Control Group: Usual Care (No Intervention): Participants will continue to receive usual outpatient or home-based rehabilitation services as recommended by their treating clinicians, including any prescribed home exercise programs. No Rise&Walk InHome device will be provided. Participants will wear an activity tracker and complete weekly logs documenting rehabilitation visits and home exercise adherence. They will also receive brief weekly remote check-in calls with the study team for clarification of step counting logs.

INTERVENTIONS:
Device: Rise&Walk InHome by Healing Innovations — The Rise&Walk InHome (RWH) is a robotic gait training technology that allows for high repetition stepping practice safely in the home. A RWH device will be placed in the homes of participants in the treatment group. If needed, refresher training will be provided upon installation, and device settings will be configured based on the participant's most recent screening session. Participants in the treatment group will be instructed to use the RWH for 30 minutes per day, four times per week. Participants can achieve 30 minutes in ≥ 10 minute bouts throughout the day or if rest breaks are needed within the session. Individualized parameters will be established at Kessler, and participants will be educated on self-progression using the RPE monitor to track effort and progress.
  Arms: Treatment Group: Rise&Walk InHome Walking Group

SUMMARY:
This pilot, parallel-group randomized controlled trial will evaluate the feasibility, safety, usability, and preliminary efficacy of the Rise&Walk InHome (RWH), a novel robotic gait training device designed for home use after stroke. Twenty adults with lower-extremity motor impairment following a first-ever stroke (3 months to 5 years post-event) will be randomized 1:1 to either (1) RWH-assisted home walking plus usual care or (2) usual care alone for 12 weeks. Participants in the intervention group will receive an in-home RWH device, complete a structured device training program, and be instructed to perform 30-minute RWH walking sessions four times per week (48 sessions total). All participants will undergo standardized outcome assessments at baseline, weeks 4, 8, and 12, including the 6-Minute Walk Test (primary outcome), 10-Meter Walk Test, daily step count via wearable activity tracker, and health-related quality of life (SF-36). Additional feasibility and usability outcomes include device use and adherence, patient satisfaction and motivation, ease of use, perceived exertion, and adverse events. Findings will inform the feasibility of in-home deployment of the RWH device and provide preliminary effect-size estimates to guide the design of a larger efficacy trial.

DETAILED DESCRIPTION:
This study is Aim 3 of a larger NIH-funded project to develop and evaluate the Rise&Walk InHome (RWH), a stationary robotic gait training device designed to deliver high-repetition, high-intensity stepping exercise in the home for individuals with walking limitations after stroke. Aims 1 and 2 focus on hardware and software usability optimization and device safety testing; Aim 3, described here, is a pilot clinical trial to assess feasibility, safety, usability, and preliminary clinical efficacy of the RWH compared with usual care.

Stroke survivors frequently face barriers to accessing clinic-based high-dose gait training, including transportation, cost, and limited availability of advanced rehabilitation technologies. High-intensity, task-specific gait training can improve walking speed, endurance, and function after stroke, yet these gains often fail to translate into increased real-world walking activity. Bringing robotic stepping into the home may improve access, enable higher cumulative training doses, and support more consistent engagement. The RWH is a transfer-accessible, body-weight-support gait trainer that transitions users from sit to stand and guides the legs through a stepping pattern while allowing adjustable body-weight offload, speed, and assistance. An integrated touchscreen interface and remote dashboard support parameter progression, safety monitoring, and adherence tracking.

This parallel-group, single-blind randomized controlled trial will enroll approximately 20 adults with a first-ever stroke and lower-extremity motor impairment who are 3 months to 5 years post-stroke and able to stand for at least 30 minutes with minimal assistance. After informed consent, eligibility screening, home evaluation, and technology competency training at the clinical site, participants will be randomized (1:1) to either the RWH intervention plus usual care or usual care alone. Randomization will occur only after participants (and, if needed, an assistant) successfully complete a structured RWH training and competency checklist and the home environment is deemed suitable for safe device installation.

Intervention group (RWH + usual care): Participants assigned to the intervention will receive an RWH device installed in their home by an engineer and physical therapist. Device settings (e.g., speed, body-weight support, assistance levels) will be individualized based on baseline assessments and in-clinic training. Participants will be instructed to perform 30-minute walking sessions on the RWH four times per week for 12 weeks (with up to 60 minutes per day allowed to accommodate warm-up, cool-down, and rest breaks). They will use the built-in Borg CR10 Rating of Perceived Exertion (RPE) tool to target high-intensity gait training during work intervals, with lower-intensity periods for recovery. Device-recorded data (session duration, step count, assistance, body-weight support, and average RPE) will be transmitted to a secure, HIPAA-compliant dashboard. Weekly phone or virtual check-ins with the study team will review progress, adjust training parameters as needed, and monitor safety and technical issues.

Control group (usual care): Participants in the control arm will continue with standard outpatient or home-based rehabilitation services as recommended by their clinical providers, including any prescribed home exercise programs. The study team will not prescribe or alter usual care. Control participants will wear a study-provided activity tracker and complete simple weekly logs to document rehabilitation visits, duration, and types of activities, as well as adherence to prescribed home exercises. Periodic check-in calls will be used to clarify logs and monitor safety.

All participants (both groups) will receive a wearable step-tracking watch to measure daily step count during a 7-day baseline period and throughout the 12-week study. Outcome assessments will be completed at baseline and at approximately 4, 8, and 12 weeks. The primary efficacy endpoint is change in walking endurance as measured by the 6-Minute Walk Test (6MWT). Secondary endpoints include walking speed (10-Meter Walk Test), daily step count, and health-related quality of life. Tertiary feasibility and usability endpoints include device adherence and total minutes of RWH use, patient satisfaction and motivation, perceived usability, session-level exertion, and qualitative feedback captured during weekly check-ins. Adverse events (AEs) and serious adverse events (SAEs) will be tracked throughout the 12-week period, classified using standard medical coding, and summarized descriptively.

The target sample size of approximately 20 participants (10 per arm) is based on feasibility considerations and will support estimation of recruitment and adherence rates, variability in key outcome measures, and preliminary between-group effect sizes. Although the trial is not powered to detect small between-group differences, it is designed to (1) determine whether in-home use of the RWH is feasible, safe, and acceptable for stroke survivors and their assistants; (2) generate preliminary effect-size estimates for changes in 6MWT, 10MWT, step counts, and quality-of-life measures; and (3) identify practical considerations for larger, multi-site efficacy trials and for future reimbursement and implementation efforts.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* First-ever ischemic or hemorrhagic stroke confirmed by medical record.
* 3 months to 5 years post-stroke at time of enrollment.
* Presence of lower-extremity motor impairment limiting walking function.
* Able to stand for at least 30 minutes with no more than minimal assistance (with or without a device).
* Medically stable and cleared by a physician to participate in moderate-intensity ambulation exercise.
* Living in a home environment that can safely accommodate device installation (e.g., adequate space, appropriate flooring, and power access) as determined by the study team.
* Able to understand study procedures and provide informed consent (or have a legally authorized representative), with sufficient cognitive and communication skills to follow simple instructions.
* If assistance is required for transfers or device set-up, availability of a caregiver or assistant willing to participate in training and device use.

Exclusion Criteria:

* Unstable cardiovascular, respiratory, or other medical conditions that contraindicate moderate- to high-intensity walking exercise (e.g., unstable angina, decompensated heart failure, uncontrolled arrhythmias).
* Severe musculoskeletal or orthopedic conditions limiting safe participation in supported stepping (e.g., unstable fractures, severe contractures preventing positioning in the device).
* Severe spasticity or movement disorders that would preclude safe use of the device, based on investigator judgment.
* Severe cognitive impairment, aphasia, or behavioral disturbance that would prevent informed consent or safe participation.
* Progressive neurological conditions (e.g., progressive neurodegenerative disease) expected to significantly worsen over the 12-week study period.
* Current participation in another interventional trial targeting gait or lower-extremity function.
* Any other condition that, in the opinion of the investigators, would make participation unsafe or interfere with study adherence or outcome interpretation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | 0,4,8,12 weeks
  A standardized submaximal exercise test that measures functional exercise capacity by recording the total distance a participant can walk on a flat, straight course in six minutes. The primary outcome is walking distance, typically recorded in meters. Higher distances indicate better functional mobility and aerobic capacity, whereas shorter distances reflect greater impairment or reduced endurance.

SECONDARY OUTCOMES:
ten-meter walk test | 0,4,8,12 weeks
  A performance-based measure of walking speed in which participants are timed while walking a 10-meter distance at their comfortable and/or fastest safe speed on a flat, level surface. Walking speed (m/s) is calculated by dividing distance in meters by time in seconds, often using the middle 6 meters to minimize acceleration and deceleration effects. Higher walking speeds indicate better functional mobility and gait performance, whereas slower speeds reflect greater gait impairment and reduced community ambulation capacity. Slower gait speeds have been associated with increased fall risk and reduced ability to safely navigate community environments.
Daily Step Count | Through study completion, on average 13 weeks.
  Cumulative change in daily step count using a Step Tracking Device
Short Form (36) Health Survey | 0,4,8,12 weeks
  A 36-item self-report questionnaire assessing health-related quality of life across eight domains: Physical Functioning, Role Limitations due to Physical Health, Bodily Pain, General Health Perceptions, Vitality (Energy/Fatigue), Social Functioning, Role Limitations due to Emotional Problems, and Mental Health. Items are scored and transformed to yield domain scores ranging from 0 to 100, with higher scores indicating better health status and quality of life (less disability/fewer limitations). Summary scores (Physical Component Summary and Mental Component Summary) may also be calculated, with higher scores reflecting better overall physical or mental health.
Modified version of the Intrinsic Motivation Inventory (IMI) designed to include 26 relevant items from the full set of 45 items in the original questionnaire. | 4,8,12 weeks
  Modified Intrinsic Motivation Inventory (IMI) for Rise&Walk InHome (RWH): An 18-item self-report questionnaire adapted from the Intrinsic Motivation Inventory to assess participants' motivation and user experience related to using the RWH device at home. Items are rated on a 7-point Likert scale (1 = Strongly Disagree to 7 = Strongly Agree). The measure includes six subscales: Interest/Enjoyment, Perceived Competence, Effort/Importance, Pressure/Tension, Value/Usefulness, and Usability & Feasibility. Pressure/Tension items are reverse-scored so that higher scores reflect lower pressure or stress. Subscale scores are calculated by summing (or averaging) the items within each domain after reverse scoring, yielding a possible range of 1-7 for each item and higher scores indicating greater intrinsic motivation, perceived competence, effort, perceived value, usability, and lower pressure/tension related to RWH use.

OTHER OUTCOMES:
Rating of Perceived Exertion (RPE) - Modified BORG | 4,8,12 weeks
  RPE will be measured for the treatment group only during their walking sessions. The technology software will use the Borg RPE scale. Responses for each domain will be rated using the revised category-ratio scale (0 [nothing at all] to 10 [maximal] ordinal response scale).
Walking compliance | 4,8,12 weeks
  e will model walking compliance as a proportion, with cumulative number of successful events from a series of successes and failures divided by the total number of assessments. The RWH system has a mobile application that shares usage data with an online HIPPA-compliant dashboard, which will be used to monitor walking compliance. Walking sessions on the RWH system will be performed 4 times per week over the course of the study. We will require a minimum of 30-minute sessions for successful participation in each walking routine.
System Usability Scale | 4,8,12 for treatment group
  Ease of use will be measured for the treatment group using the System Usability Scale (SUS). Each of the 10 questions on the SUS will be answered on a 5 pt ordinal scale, with responses ranging from "strongly agree" to "strongly disagree". The final possible scores ranging from 0 to 40 will be transformed to a 0 to 100 scale, based on the assumption that each question carries equal weight.
Cumulative incidence of adverse events | Through Study Completion, approximately 12 months
  Adverse events (AEs) will be classified according to the International Classification of Diseases Version 10 (ICD-10) or another validated coding system for medical complications. Individual AE types will also be summarized.
Cumulative incidence of treatment-related and serious adverse events | Through Study completion, approximately 12 months
  An AE is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes: a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Incidence of SAEs will be monitored until final follow-up or upon study exit.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Hartman, DPT, Principal Investigator — Healing Innovations; Karen Nolan, PhD, Principal Investigator — Kessler Foundation; Ben Taylor, Principal Investigator — Healing Innovations
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hornby TG, Reisman DS, Ward IG, Scheets PL, Miller A, Haddad D, Fox EJ, Fritz NE, Hawkins K, Henderson CE, Hendron KL, Holleran CL, Lynskey JE, Walter A; and the Locomotor CPG Appraisal Team. Clinical Practice Guideline to Improve Locomotor Function Following Chronic Stroke, Incomplete Spinal Cord Injury, and Brain Injury. J Neurol Phys Ther. 2020 Jan;44(1):49-100. doi: 10.1097/NPT.0000000000000303. PMID 31834165
- [Background] Mehrholz J, Thomas S, Kugler J, Pohl M, Elsner B. Electromechanical-assisted training for walking after stroke. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD006185. doi: 10.1002/14651858.CD006185.pub5. PMID 33091160
- [Background] Luo L, Zhu S, Shi L, Wang P, Li M, Yuan S. High Intensity Exercise for Walking Competency in Individuals with Stroke: A Systematic Review and Meta-Analysis. J Stroke Cerebrovasc Dis. 2019 Dec;28(12):104414. doi: 10.1016/j.jstrokecerebrovasdis.2019.104414. Epub 2019 Sep 27. PMID 31570262
- [Background] de Menezes KKP, Ada L, Teixeira-Salmela LF, Scianni AA, Avelino PR, Faria CDCM, Nascimento LR. Home-Based Interventions may Increase Recruitment, Adherence, and Measurement of outcomes in Clinical Trials of Stroke Rehabilitation. J Stroke Cerebrovasc Dis. 2021 Oct;30(10):106022. doi: 10.1016/j.jstrokecerebrovasdis.2021.106022. Epub 2021 Aug 4. PMID 34364011
- [Background] Hu MM, Wang S, Wu CQ, Li KP, Geng ZH, Xu GH, Dong L. Efficacy of robot-assisted gait training on lower extremity function in subacute stroke patients: a systematic review and meta-analysis. J Neuroeng Rehabil. 2024 Sep 19;21(1):165. doi: 10.1186/s12984-024-01463-1. PMID 39300491